CLINICAL TRIAL: NCT06918938
Title: Unraveling Visuomotor Control in Parkinson Disease With and Without Freezing of Gait
Brief Title: Visuomotor Control in Parkinson Disease
Status: Recruiting | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202502008RINB
Record Dates: First submitted 2025-03-27; First posted 2025-04-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease; Transcranial magnetic stimulation; Motor control
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- FOG: Participants with Parkinson disease and freezing of gait
- NFOG: Participants with Parkinson disease without freezing of gait
- CON: Age-matched healthy adults

SUMMARY:
Visuomotor processing is the ability to integrate visual information into motor plans and movement correction, which is highly required in daily activities such as writing and walking. As visual impairments have been reported in people with Parkinson's disease (PD), it is likely that those impairments may affect visuomotor processing ability and subsequently impair motor performance. Furthermore, people with PD and freezing of gait (FOG) have exhibited poorer visual perception than those without FOG, yet the differences of visuomotor control have not been well investigated. Additionally, little did the studies apply neurophysiological assessment to investigate the associated neural mechanisms. This study aims to investigate behavioral and neurophysiological differences in visuomotor control among people with PD and FOG (freezers), without FOG (non-freezers), and age-matched healthy controls. Sixty-three participants, 21 freezers, 21 non-freezers, and 21 age-matched healthy controls, will be enrolled in this study. Behavioral assessments, including a manual control task and visual perception tests will be used to evaluate visuomotor and visual perceptual abilities. Neurophysiological correlates, including corticomotor excitability and corticocortical connectivity between V1-M1 and PPC-M1, will be examined using transcranial magnetic stimulation. It is hypothesized that freezers will demonstrate the greatest visuomotor impairments and disrupted corticocortical connectivity compared to non-freezers and controls. By integrating behavioral and neurophysiological outcomes, this study seeks to unravel the mechanisms linking visual and motor impairments to FOG, ultimately providing insights into targeted interventions to improve visuomotor processing and motor performance in PD.

ELIGIBILITY:
Inclusion Criteria:

* age above 18
* able to follow the researchers' instructions
* normal or correct-to-normal vision to view a computer screen

Exclusion Criteria:

* neurological disorders other than PD
* diagnosed psychological disorders or a tendency of anxiety and/or depression
* a self-history of seizure or a family history of epilepsy
* deep brain stimulation or pacemaker implanted
* unstable cardiovascular diseases or other uncontrolled medical conditions
* pregnant
* surgical history, severe injury, or severe tremor of their upper extremities that can affect their movements in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with PD are idiopathic PD diagnosed by a neurologist, while healthy controls are absent of any neurological disorders.
Sampling Method: Probability Sample
Enrollment: 63 (Estimated)
Dates: Start 2025-07-19 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Root-mean square-error | Day 1
  Overall performance accuracy relative to the target waveform, which is the mean difference between the target waveform and the participant's movement trajectory calculated over their actual movement time.
Directional error | Day 1
  The value of the instantaneous component of the hand movement vector, perpendicular to the target trajectory in every sampled time point, which will be calculated and expressed as a percentage of the total movement vector
Squared mean jerk | Day 1
  The squared mean of the jerk of the visuomotor trajectory, which a minor JSM is assumed a major smoothness by better controlling the movement.
Movement time | Day 1
  Total movement time of a trial will be recorded.
Tracking interruption | Day 1
  Frequency and duration of tracking interruptions will be recorded when the participant's cursor exits the target circle.

SECONDARY OUTCOMES:
Benton Judgment of Line Orientation Test | Day 2
  A 30-item neuropsychological assessment of visuospatial ability. Participants are required to match 2 angled line portions on the top page to an array of 11 target lines, and the correction rate will be recorded.
Random dot cinematogram | Day 2
  A psychological assessment of visual motor perception. Participants need to distinguish the coherent motion direction, and the correction rate and minimal detectable threshold of coherence will be recorded.
National Eye Institute Visual Function Questionnaire-25 | Day 2
  A 25-item self-reported questionnaire of visual-related activities, which the total score will be recorded.
Purdue Pegboard Test | Day 2
  A behavioral assessment of hand dexterity ability. Participants are instructed to use one or both hands to sequentially move as many pegs into two parallel rows of holes as possible, within a set time limit, and the movement time will be recorded.
Timed Up and Go Test | Day 2
  A behavioral assessment of dynamic balance ability. Participants will be instructed to rise from a chair, walk for 3 meters, turn around, return to the chair, and sit down, and the movement time will be recorded.
Movement Disorder Society Unified Parkinson's Disease Rating Scale | Day 1
  A comprehensive scale of Parkinson disease characteristics, including non-motor aspects of experiences of daily living, motor aspects of experiences of daily living, motor examination, and motor complications. Scores of each subscales will be recorded.
New Freezing of Gait Questionnaire | Day 1
  A self-reported questionnaire to evaluate the frequency and severity of freezing of gait in people with PD, which the total score will be recorded.
Cortical excitability | Day 1 and Day 2
  Transcranial magnetic stimulation (TMS) device (The Magstim Company Ltd, Whitland, UK) will be used to determine the neurophysiology of corticomotor excitability.
Corticocortical connectivity | Day 1 and Day 2
  Transcranial magnetic stimulation (TMS) device (The Magstim Company Ltd, Whitland, UK) will be used to determine the neurophysiology of corticocortical connectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Graduate Institute of Physical Therapy, Principal Investigator — National Taiwan University
Locations (1):
- School and Graduate Institute of Physical Therapy, Taipei, Zhongzheng Dist., Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Inzelberg R, Schechtman E, Hocherman S. Visuo-motor coordination deficits and motor impairments in Parkinson's disease. PLoS One. 2008;3(11):e3663. doi: 10.1371/journal.pone.0003663. Epub 2008 Nov 6. PMID 18987752
- [Background] Palomar FJ, Conde V, Carrillo F, Fernandez-del-Olmo M, Koch G, Mir P. Parieto-motor functional connectivity is impaired in Parkinson's disease. Brain Stimul. 2013 Mar;6(2):147-54. doi: 10.1016/j.brs.2012.03.017. Epub 2012 Apr 15. PMID 22537863